CLINICAL TRIAL: NCT04993313
Title: A Randomized Trial of Standard Verbal Counseling With or Without a Pictorial Educational Tool to Reduce Psychological Morbidity in Women Receiving Breast Radiation Therapy
Brief Title: Standard Verbal Counseling With or Without a Pictorial Educational Tool for the Reduction of Psychological Morbidity in Patients With Stage 0-IIIA Breast Cancer Receiving Radiation Therapy, COPE Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Carl Post, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00020501; NCI-2021-06325 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00020501 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2021-07-09; First posted 2021-08-06 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Anatomic Stage 0 Breast Cancer AJCC v8; Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage 0 Breast Cancer AJCC v8; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Breast Carcinoma
MeSH Terms: conditions — Breast Carcinoma In Situ; Breast Neoplasms | interventions — Counseling; Early Intervention, Educational; Educational Status; Methods; Surveys and Questionnaires

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (counseling, photo guide) (Experimental): Patients undergo verbal counseling and view a photo guide. Patients also complete questionnaires at 2 weeks, 6 and 12 months.
  Interventions: Other: Counseling; Other: Educational Intervention; Behavioral: Questionnaire
- Arm II (counseling) (Active Comparator): Patients undergo verbal counseling. Patients also complete questionnaires at 2 weeks, 6 and 12 months.
  Interventions: Other: Counseling; Behavioral: Questionnaire

INTERVENTIONS:
Other: Counseling — Undergo verbal counseling
  Other Names: Counseling Intervention
Other: Educational Intervention — View photo guide
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm I (counseling, photo guide)
Behavioral: Questionnaire — Complete questionnaires
  Other Names: Questionnaires

SUMMARY:
This clinical trial studies the effect of standard verbal counseling with or without a pictorial educational tool for the reduction of psychological morbidity in patients with stage 0-IIIA breast cancer receiving radiation therapy. Beginning radiation therapy for breast cancer can be stressful. Education about what to expect often reduces the stress, anxiety, and depression experienced by these patients. This study is being done to see how effective photos are in reducing stress, anxiety, and depression associated with radiation therapy for patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assessment of patient reported anxiety and depression, confidence with information, and side effect expectations of radiation therapy following counseling with or without photo guide at pre-treatment, 2 weeks, 6 months, and 12 months.

SECONDARY OBJECTIVE:

I. Efficacy of intervention to impart reasonable expectations of the side effect burden of radiation therapy (RT).

EXPLORATORY OBJECTIVE:

I. Picture Guide book.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo verbal counseling and view a photo guide. Patients also complete questionnaires at 2 weeks, 6 and 12 months.

ARM II: Patients undergo verbal counseling. Patients also complete questionnaires at 2 weeks, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients diagnosed with stage 0-IIIA disease who are planned to receive adjuvant hypofractionated or standard fractionated radiation treatment
* Patients must have the ability to read and understand English

Exclusion Criteria:

* Patients who are planned for ultra-hypofractionated radiation treatment
* Patients who are planned for partial breast radiation treatment
* Patients who are planned to receive concurrent radiosensitizing chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in patient reported anxiety and depression | Baseline to 12 months
  Will use items from the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (CTCAE). Depression and anxiety will be analyzed as binary outcomes. Will compare questionnaire scores for anxiety and depression between the two groups. Scores will be reported as descriptive using CTCAE grading scale ranging from "mild" (1) to "life threatening" (4).

SECONDARY OUTCOMES:
Cosmesis expectations versus self-reported experiences | Up to 12 months
  Assessed through a custom survey.

OTHER OUTCOMES:
Accurate knowledge of radiation therapy side effects | Up to 12 months
  Assessed through a custom survey. This will be assessed using a custom questionnaire that assesses the patient's perception of their own understanding of radiation-related side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Carl Post, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification, will be shared with anyone who wishes to access the data following a request proposal. Types of analyses included will be based on the approved proposal.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Proposals should be directed to xxx@yyy. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link: https://www.ohsu.edu/octri/redcap-your-complete-solution-online-databases-and-surveys-research)